CLINICAL TRIAL: NCT00365612
Title: Phase IV, Open-Label, Randomized, Multicenter Study Evaluating Efficacy and Tolerability of Single Tablet Regimen of Efavirenz/Emtricitabine/Tenofovir DF Compared to Unmodified HAART in HIV-1 Infected Subjects Who Have Achieved Virological Suppression on Their HAART Regimen
Brief Title: Single Tablet Regimen (STR) Simplification Study for HIV-1 Infected Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: John Flaherty, Director, Medical Affairs, Gilead Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AI266073
Record Dates: First submitted 2006-08-16; First posted 2006-08-17 (Estimated); Last update posted 2008-04-10 (Estimated); Status verified 2008-04

CONDITIONS: HIV Infections
Keywords: HIV; HIV-1; AIDS; Human Immunodeficiency Virus; HIV-1 Infection
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — efavirenz; Emtricitabine; Racivir; Tenofovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Efavirenz (EFV), Emtricitabine (FTC), Tenofovir DF (TDF)

SUMMARY:
To compare the effectiveness (efficacy, safety & tolerability) of a Single Tablet Regimen of efavirenz/emtricitabine/tenofovir DF to subjects continuing on unmodified HAART as measured by the proportion of patients who maintain viral load (HIV-1 RNA) <200 copies/mL at Week 48.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 positive patients who have maintained an HIV-1 viral load <200 copies/mL, for at least 3 months.
* Patients must be on their first HAART or have documented viral suppression on a PI-based regimen at the time of any prior change in therapy.
* HAART must consist of either:

  1. A PI (with or without ritonavir) + at least 2 NRTIs or
  2. An NNRTI + at least 2 NRTIs.
* Negative serum pregnancy test.

Exclusion Criteria:

* Patients who have taken any NNRTI prior to their current therapy.
* Patients who have taken a NRTI-only therapy for greater than 7 days prior to their current therapy.
* Patients who are currently taking EFV+FTC+TDF.
* Patients who have a creatinine clearance of <60 mL/min by Cockcroft-Gault estimation.
* Patients who have experienced virologic failure with any previous ARV therapy.
* Patients who have documented resistance to any of the study agents at any time in the past.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2006-07; Primary Completion 2007-10 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Primary: Proportion of patients with HIV-1 RNA levels <200 copies/mL at Week 48
Safety Outcome Measures: Adverse Events, Laboratory Tests
Outcomes Research Measures: Quality of life, adherence, preference of medication, perceived ease of regimen, HIV symptoms

CONTACTS AND LOCATIONS:
Overall Officials: John Flaherty, Study Director — Gilead Sciences
Locations (55):
- United States (53):
  - Hobson City, Alabama
  - Phoenix, Arizona
  - Beverly Hills, California
  - Long Beach, California
  - Los Angeles, California
  - Oakland, California
  - San Diego, California
  - San Francisco, California
  - Tarzana, California
  - Denver, Colorado
  - Norwalk, Connecticut
  - Washington D.C., District of Columbia
  - Fort Lauderdale, Florida
  - Hollywood, Florida
  - Miami, Florida
  - Orlando, Florida
  - Pensacola, Florida
  - Port Saint Lucie, Florida
  - Safety Harbor, Florida
  - Tampa, Florida
  - Vero Beach, Florida
  - Atlanta, Georgia
  - Decatur, Georgia
  - Aurora, Illinois
  - Chicago, Illinois
  - Indianapolis, Indiana
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Springfield, Massachusetts
  - Berkley, Michigan
  - Grosse Pointe Woods, Michigan
  - Minneapolis, Minnesota
  - St Louis, Missouri
  - Hillsborough, New Jersey
  - Newark, New Jersey
  - Somers Point, New Jersey
  - Albany, New York
  - Brooklyn, New York
  - Mount Vernon, New York
  - New York, New York
  - Rochester, New York
  - Charlotte, North Carolina
  - Greenville, North Carolina
  - Winston-Salem, North Carolina
  - Akron, Ohio
  - Philadelphia, Pennsylvania
  - Providence, Rhode Island
  - Dallas, Texas
  - Harlingen, Texas
  - Houston, Texas
  - Annandale, Virginia
  - Hampton, Virginia
  - Spokane, Washington
- Puerto Rico (2):
  - Ponce
  - San Juan

REFERENCES:
- [Derived] Hodder SL, Mounzer K, Dejesus E, Ebrahimi R, Grimm K, Esker S, Ecker J, Farajallah A, Flaherty JF; AI266073 Study Group. Patient-reported outcomes in virologically suppressed, HIV-1-Infected subjects after switching to a simplified, single-tablet regimen of efavirenz, emtricitabine, and tenofovir DF. AIDS Patient Care STDS. 2010 Feb;24(2):87-96. doi: 10.1089/apc.2009.0259. PMID 20156091
- [Derived] Dejesus E, Young B, Morales-Ramirez JO, Sloan L, Ward DJ, Flaherty JF, Ebrahimi R, Maa JF, Reilly K, Ecker J, McColl D, Seekins D, Farajallah A; AI266073 Study Group. Simplification of antiretroviral therapy to a single-tablet regimen consisting of efavirenz, emtricitabine, and tenofovir disoproxil fumarate versus unmodified antiretroviral therapy in virologically suppressed HIV-1-infected patients. J Acquir Immune Defic Syndr. 2009 Jun 1;51(2):163-74. doi: 10.1097/QAI.0b013e3181a572cf. PMID 19357529
- See also: ATRIPLA website — http://www.atripla.com
- See also: Gilead Sciences website — http://www.Gilead.com
- See also: Bristol-Myers Squibb website — http://www.BMS.com